CLINICAL TRIAL: NCT00091767
Title: Genetic Studies in Difficult to Treat Asthma: TENOR
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1270; R01HL076285-03 (NIH)
Record Dates: First submitted 2004-09-16; First posted 2004-09-20 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2008-07

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To investigate genetic factors that affect asthma severity.

DETAILED DESCRIPTION:
BACKGROUND:

The TENOR (The Epidemiology and Natural History of Asthma: Outcomes and Treatment Regimens) study is an ongoing three-year multi-center observational cohort study of 4756 severe or difficult-to-treat patients with asthma aged 6 or older. Of this group of asthmatics, 44.6% meet the National Heart, Lung, and Blood Institute National Asthma Education and Prevention Program guidelines for severe persistent asthma, 27.5% for moderate persistent asthma, and 27.8% for mild persistent asthma. All subjects were evaluated initially with comprehensive questionnaires and laboratory testing, and are then seen every 6 months during the remaining 3 years of the study. Phenotypic information collected includes information on asthma exacerbations, medication use, urgent care visits, quality of life, pulmonary function tests (spirometry with reversibility), total serum IgE levels, and history of allergies. If accessed now, before the termination of the TENOR study, this population represents one of the largest populations of phenotypically characterized difficult-to-treat and severe asthmatics potentially available for genomic and pharmacogenetic studies. TENOR will finish at the end of 2004, thus there is a very short time window in which to obtain DNA samples for genetic studies before the termination of the study. Isolation and storage of DNA from this well characterized, longitudinal population will serve as a resource not only for the studies in this grant but also for future genomics and pharmacogenetic studies in asthma.

DESIGN NARRATIVE:

The study investigates genetic factors that affect asthma severity in the TENOR subjects. The study tests the hypothesis that factors which produce difficult-to-treat and severe asthma are produced by altered inflammatory responses that are related, at least in part, to sequence variants (polymorphisms) in genes that regulate inflammation, allergic responsiveness, and/or affect structural components in the airways. The study also tests the hypothesis that some patients develop more severe asthma because of genetic differences that modulate their responses to pharmacologic agents. To test these hypotheses, the following specific aims will be carried out: 1) Obtain DNA samples from at least 4,000 asthmatics currently enrolled in the ongoing TENOR study; 2) Determine whether sequence variants (polymorphisms) in genes that regulate inflammation, cellular responses, and/or tissue injury and repair are more frequently associated with asthma severity using the baseline data; 3) Determine the importance of genetic polymorphisms in genes that may be important in IgE regulation in this population of difficult-to-treat patients with asthma; 4) Evaluate pharmacogenetic relationships between polymorphisms in the a2 adrenergic receptor (a2AR) in those subjects on long-acting beta-2-agonists to determine the effect on asthma severity; 5) Evaluate pharmacologic mechanisms by investigating whether polymorphisms in genes that regulate responses to asthma therapy are more frequent in severe disease.

ELIGIBILITY:
No eligibility criteria

Ages: 6 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Bleecker — Wake Forest University Health Sciences